CLINICAL TRIAL: NCT01261221
Title: Pilot Study of Metabolic Syndromes and HIV Infections in Indian Tibetans
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUH-IRB-990168
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2011-07

CONDITIONS: Metabolic Syndromes; HIV Infection
MeSH Terms: conditions — Metabolic Syndrome; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Kaohsiung Medical University Chung-Ho Memorial Hospital will provide a long-term free medical service in Indian Tibetans since July 2010. The investigators plan to investigate metabolic syndromes and HIV infection in Indian Tibetan community. The investigators will survey the prevalence and risk factors by means of HIV quick test and questionnaires. Since there is lacking of prevalence survey for metabolic syndrome and HIV infection in Tibetan colony of India, the investigiators will carry out this survey under the support and assistance of Department of Health of Central Tibetan Government.

ELIGIBILITY:
Inclusion Criteria:

Tibetan colony of India

Exclusion Criteria:

non-Tibetan colony of India

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Tibetan colony of India
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung, Taiwan